CLINICAL TRIAL: NCT03221413
Title: A Translational, Multimodal Approach to Implementing Non-invasive Paradigms for the Treatment of Oscillopathies
Brief Title: Transcranial Alternating Current for Oscillopathies
Acronym: tACS_EEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UPadova
Record Dates: First submitted 2016-02-11; First posted 2017-07-18 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2019-08

CONDITIONS: Parkinson Disease; Pain
Keywords: transcranial alternating current stimulation; Neuroimaging; EEG
MeSH Terms: conditions — Parkinson Disease; Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- PD tACS (Experimental): Persons with Parkinson disease who will be treated with tACS: Intervention: tACS (transcranial alternating current stimulation)
  Interventions: Device: transcranial alternating current stimulation (tACS)
- Pain tACS (Experimental): Persons with neuropathic pain who will treated with tCAS. Intervention: tACS (transcranial alternating current stimulation)
  Interventions: Device: transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: transcranial alternating current stimulation (tACS)

SUMMARY:
The need for non-invasive, non-pharmacological and cost-effective therapeutic options has revived the use of transcranial current stimulation, either direct (tDCS) or alternating (tACS), in a wide range of pathologies and cognitive disturbances. Results, although often promising, are not unequivocal, possibly due to different stimulation parameters and sites, or non-homogenous patient selection. tDCS has been widely applied but few studies have focused on tACS which has the advantage of potentially entraining brain oscillations at the same frequency of stimulation. This overcomes the basic mechanism of tDCS which deploys anodal or cathodal currents to broadly excite or inhibit supposedly dysfunctional underlying cortex.

Whether a stimulation paradigm based on sound neurophysiological markers could provide a better and longer-lasting clinical outcome has not yet been ascertained.

The investigators aim to establish, with a trans-disease approach, categories characterized by defective EEG oscillatory activity and related dysfunctional networks. This classification, expected as the result of the first stage of this project, will guide the stimulation paradigm: categories with a pathologically low-band EEG prevalence will be treated with high-frequency tACS, and vice-versa, while the stimulation site will correspond to the defective sites of pathological EEG band maps. Parkinson's disease (PD), the EEG marker of which is a shift towards fast frequencies, and neuropathic pain (NP), with an EEG prevalence of slow bands, will be considered.

In order to categorize pathologies on the basis of their EEG frequencies, EEG power spectrums will be derived from resting EEG, and cortical oscillatory reactivity will be assessed by EEG-TMS (electroencephalographic-Transcranial Magnetic Stimulation) co-registration. This method appears to elicit state-dependent brain oscillatory response and is expected to support power spectrum data. The identified prevailing EEG band will be used subsequently to reconstruct scalp EEG band distribution. tACS paradigms will be tailored according to these findings: the anode will be placed over the scalp area corresponding to the dysfunctional rhythm and frequency will be set in order to correct the prevailing EEG band (slow stimulation if fast frequencies prevail, and vice-versa).

The translational element of this research proposal will consist of its clinical application in day-to-day practice for the benefit of people with the target conditions. The patient-groups, after undergoing the neurophysiology studies, will be tested with disease-specific scales and a neuropsychological battery. A 2-weeks tACS, either real or active sham, protocol will then be performed (30 minutes/day, 5 days/week), associated with an ad hoc rehabilitation protocol (60 minutes/day 5 days/week). During the last day of stimulation, patients will be tested again with the disease specific scales, neuropsychological battery and standard EEG to detect EEG frequencies modifications. At 4-weeks follow up, the same tests and EEG recording will be carried out, to assess the persistence of after-effects.

The expected result is a valid, non-invasive and cost-effective stimulation paradigm based on sound neurophysiologic markers which transcend traditional disease classifications.

DETAILED DESCRIPTION:
tDCS has been applied to a spectrum of diseases, including depression, Parkinson's disease (PD), dementia and others, on the basis of the concept of dysfunctional brain areas: modulating the hypo-or hyper-function of the indicated brain regions via anodal or cathodal tDCS has shown evidence of clinical symptom improvement, although generally short lasting and often with discordant results among studies. Conversely, tACS has only rarely been applied to people with disease, with discordant results. Its application to healthy individuals to boost sleep and sleep-related memory formation and working memory has, however, been shown to be effective. If consensus on stimulation patterns (continuous vs. alternating) is, however, lacking, the same holds true for frequencies, although evidence from computational and animal studies demonstrates that tACS is very effective at entraining the network at the frequency of the applied stimulation, with theta noticeably efficacious at improving cognitive performances in memory tasks.

Whether a different paradigm, tailored to specific neurophysiological signatures, and not to the phenotype of the underlying dysfunction (i.e. applying inhibitory tDCS on the hyperfunctioning cortical area of a given disease or vice-versa), could lead to better and long-lasting clinical results is not yet defined.

Therefore, this proposed study has two fundamental questions: 1) is a re-categorization of pathologies based on their oscillatory activities and related scalp distribution. Indeed, the answer the investigators are seeking is whether the investigators could identify clear neurophysiological markers that could lead to a new diagnostic classification. From a translational perspective the question is: 2) could these markers eventually guide therapeutic options? If these points are proved, the investigators expect to expand the results to other oscillopathies (i.e. schizophrenia or insomnia).

The objective of this project is thus two-staged: a first stage will define neurophysiologic markers of diverse diseases, overcoming the traditional symptom-based classification of pathologies. In the second stage, these features will be translated into a tailored non-invasive brain stimulation (NIBS) protocol. Indeed, focusing on oscillatory rhythms dysfunctions, tACS, that entrains specific EEG frequencies, instead of tDCS, that hypo-hyperpolarizes indiscriminately vast brain regions, will be applied.

In the first stage, selected pathologies among the broader spectrum of thalamo-cortical-dysrhythmias (TCDs) will be categorized on the basis of their prevalent EEG rhythm; in addition, oscillatory brain response to external perturbation (frequency bands synchronization or desynchronization in response to TMS stimulation as defined by EEG-TMS co-registration) will be obtained. The identified EEG frequency will subsequently be extracted from EEG to visualize scalp defective areas. The investigators will identify:

* the prevailing EEG rhythm in a resting, standard EEG by means of power spectral analysis, based on Fourier transform;
* a more detailed insight into brain reactivity and its oscillatory response as a reaction to random, non-entraining TMS stimulation with EEG co-registration, a method that appears to elicit state-dependent brain oscillatory response; Pathologies presenting with analogous neurophysiological signatures will be grouped together in order to define an appropriate, common stimulation paradigm, independently of symptom phenotype.

In the second stage the investigators will attempt to tailor tACS on the basis of the previously defined categories. The scalp area of the dysfunctional rhythm will aid in the selection of the stimulation site, whereas the stimulation paradigm will be established on the basis of the prevailing EEG bands at rest and after perturbation - i.e. transcranial stimulation will be low frequency (4 Hz) alternating (tACS) for diseases characterized by a pathological increase of fast rhythms, and vice-versa (30 Hz), in order to entrain the defective EEG band. A clear-cut, long-lasting improvement of clinical symptoms is expected.

Our expected result is to be able to set up appropriate and effective tACS stimulation paradigms based on disease neurophysiological markers rather than on clinical symptoms. Given the large number of pathologies encompassed in the TCD spectrum, this therapeutic option could become a promising non-invasive, cost-effective therapeutic option with a wide field of applications.

Pathologies to be included are:

* PD: altered thalamo-cortical loop that reflects, through the thalamus, the beta prevalence in the deep nuclei loop and reverberates to the cortex.
* Neuropathic pain (NP): evidence of increased high theta band power (7-8Hz), especially over frontal and somatosensory cortex. The generation of low-frequency activity by the thalamocortical circuit results in a long-term pathological equilibrium in the cortical pain matrix.

  2 - Methods

2.1. Pre- (T0), post-stimulation (T1) and 4weeks follow-up (T2) clinical assessment

* PD: UPDRS III, Dynamic Gait Index
* NP: Neuropathic Pain Questionnaire (NPQ), VAS for pain, Short Form 36-item Health Survey (SF-36) Possible therapy modification dictated by the individual's clinical status will be recorded.

2.2. T0, T1 and T2 neuropsychological assessment All patient groups will undergo the following neuropsychological tests battery. Anxiety state and trait will be measured and BDI administered.

* Montreal Cognitive Assessment (MoCA)
* State-Trait Anxiety Inventory (STAY) Y1 e Y2
* Beck Depression Inventory (BDI) II
* Rey Auditory Verbal Learning Test
* Rey-Osterrieth Complex Figure Test version I and III
* Modified Taylor Test
* Geriatric depression scale (short form)
* Cifrario
* Phonemic fluency test
* Edinburgh handedness Test
* Short-form Intelligence Test (TIB)
* Hopkins Verbal learning test revised (HVLTR)
* Trail making test

2.3. Signal analysis T0, T1 and T2 resting EEG analysis. EEG will be acquired using an TMS compatible EEG amplifier (BrainAmp 32MRplus, BrainProducts GmbH, Munich, Germany) and a cap providing 30 Ag/AgCl electrodes positioned according to a 10/20 system. Data will be processed in Matlab (MathWorks, Natick, MA) using scripts based on EEGLAB (http://www.sccn.ucsd.edu/eeglab), as well as a dedicated home-made code created for this study. Visible artifacts in the EEG will be removed using an independent component analysis procedure and EEG will be band-pass filtered from 1 to 30 Hz. EEG data will be divided into epochs of 2 s and a fast Fourier transform (FFT) will be applied to non-overlapping epochs, and averaged across epochs. Based on power spectra density, relative powers (%) in delta (1-4 Hz), theta (4-7Hz), alpha (8-12 Hz), and beta (13-30 Hz) frequency ranges will be evaluated.

A one sample z-test will be applied to compare the map of the patient to the grand average of the controls (a group of 20 healthy subjects). Thus, the statistical map defines the sensors in which relative power from an individual patient differs statistically from that of a reference population (control group).

Pre-stimulation (T0) EEG-TMS co-registration TMS will be performed using a Dymeg in biphasic pulse configuration (DuoMag, EMS, Italy) which generates a maximum magnetic field of 1.5 T. TMS will be delivered through a figure-of-eight focal coil over the dominant primary motor area (M1). Motor evoked potentials (MEPs) will be recorded from the left/right thenar eminence muscle with Ag/AgCl surface electrodes fixed to the skin with a belly-tendon montage. Stimulus intensity will be set at 110% of motor threshold intensity. 100 TMS single-pulse stimuli will be delivered at random, with inter-trial interval between 8-15 s.

EEG will be acquired using the same magnetic resonance compatible EEG system previously described. EEG data will be analysed using a time-frequency procedure to characterize TMS-induced oscillations. Time-frequency analysis will be performed with continuous Morlet wavelet transform, which provides a time course after magnetic stimulation of the relative power in the main frequency bands, as described above. Profiles for each subject will be averaged from the post-stimulus trials and normalized to the baseline value.

2.4. TADCS stimulation paradigm Stimulation will be applied by a battery driven external stimulator (BrainStim, EMS, Bologna, Italy) via two sponge electrodes (5x7cm). The anodal electrode will be placed over the scalp area corresponding to the defective network node as derived by EEG source analysis. The cathodal electrode will be placed over the ipsilateral mastoid. A sinusoidal current, ranging from 1 to 2mA will be delivered; stimulation frequency will be derived from the defective EEG band - i.e. if low frequency oscillations prevail, stimulation will be at 30 Hz; if high frequency oscillations prevail, stimulation will be at 4 Hz. Sham stimulation, according to consensus statement, will be delivered as random noise stimulation (RNS) with electrodes located at the same sites as active stimulation and Sham Sessions will last 30 minutes, and repeated for two weeks on 5 consecutive days per week separated by a 2 days interval. A random Noise Stimulation (RNS) with an amplitude 1 to 2 mA will be applied.

2.5. Ethical Committee Approval The study involves stimulation of human subjects and as such will require Ethical approval. The investigators obtained Ethical Approval from the Ethics Committee of the University Hospital, Padova (3507/15).

2.6. Statistical analysis and study power Data will be summarized using descriptive statistics. Appropriated 95% confidence intervals (CIs) for each outcome will be produced.

2.6.1. First phase The proportion of people with PD displaying EEG beta peak (FFT) and the 95% binomial CI will be computed. The same analysis will be performed for people with NP displaying EEG theta peak (FFT).

2.6.2. Second phase 2.6.2.1. Primary analyses A repeated measures test (ANCOVA) will be used to evaluate differences in UPDRS score and NPQ score between T0 and T1.

2.6.2.2. Secondary analyses Cross sectional evaluation at pre- and post-treatment between PD with beta Peak and PD with other EEG peaks will be run using the independent sample t test. Same analysis will be performed to evaluate differences at T0 and T1 between NP subjects with theta Peak vs NP with other EEG peaks.

Further analyses could be performed using analysis of variance (ANOCOVA) to account for these predictors: age, sex, disease severity at T0, interaction with other frequency bands, pre- and post-stimulation therapy after real and active sham tACS modification, drugs. Repeated measures models could be used.

2.6.3. Signal analysis

Analysis of variance (ANOVA) for repeated measures will be applied to the relative power with the factor ''time'' (T0, T1 and T2); the sphericity assumption will be assessed using Mauchly's test. Greenhouse-Geisser epsilon adjustments for non-sphericity will be applied where appropriate. A post hoc paired sample two tailed t-test adjusted for multiple comparisons with the Bonferroni method will be used. Statistical significance will be set at p < 0.05, corrected. Two-dimensional grand mean t-maps of the relative power will be computed from the t-values to check the topographical distribution of the significance.

2.6.4. Study power To compute the total sample size of the project the investigators will first compute the sample size for phase II. Given sample size for phase II, sample size for phase I will be computed accounting for potential drop-outs.

Phase II sample size Two different populations will be investigated (PD, NP) hence no correction for multiplicity will be performed.

People with PD and NP A sample size of 15 achieves 92% power to detect a mean of paired differences (UPDRS pre- and post-stimulation score difference) of 4.0 with an estimated standard deviation of differences of 4.3 and with significance level (alpha) of 0.05 using a two-sided paired t-test in people with PD displaying EEG beta (FFT). The same assumption will be assumed for NPQ decrease, hence a total of 30 subjects will be required, 15 for each category.

Phase I sample size The investigators expect all people with PD to have a beta frequency peak, while those with NP will be in the theta band. A sample size of 15 people with NP produces a one sided 97.5 binomial CI of 79.61%-100% given that the expected proportion of theta is 100%. A sample size of 15 people with PD produces a one sided 97.5 binomial CI of 79.61%-100% given that the expected proportion of beta is 100%.

Total sample size In order to account for potential drop outs the investigators will recruit 20 people with NP and 20 people with PD, giving a total sample size of 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* PD: diagnosis of idiopathic PD within the last 5 years (UK Brain Bank criteria); stable dose of antiparkinson therapy for at least 4 weeks; total off-medication motor Hoen and Yahr 1-2.
* NP: stable chronic pain for at least the preceding six months; score greater than or equal to 3 (0 no pain, 10 worst pain) on the visual analog scale (VAS) for pain perception during the last month before start of stimulation; refractoriness to drugs for pain relief (pain resistance to at least two of these drugs supplied in adequate dosages for 6 months).

Exclusion Criteria:

* PD: concomitant psychiatric disorder; benzodiazepine treatment; Mini Mental State Examination (MMSE) <26
* NP: clinically significant or unstable medical or psychiatric disorder, history of substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of people displaying fast brain oscillatory activity [measured as electroencephalographic (EEG) beta band prevalence] | 1 year (first)
  EEG power spectral maps will identify this category
Proportion of people dispalying slow brain oscillatory activity [measured as electroencephalographic (EEG) theta band prevalence] | 1 year (first)
  EEG power spectral maps will identify this category
Improvement ≥ 30% of the total off-medication on a motor performance scale (Unified Parkinson's Disease Rating Scale,part III) | 1 to 2 years (2nd year)
  UPDRS III is a scale measures motor preformance specifically in Parkinson's Disease
Pain reduction, measured with a specific scale (NPQ-Neuropathic Pain Questionnaire), as a reduction of at least 4 points | 1 to 2 years (2nd year)
  NPQ (Neuropathic Pain Questionnaire) is a scale measures pain

SECONDARY OUTCOMES:
Modifications of frequencies of oscillatory brain activity, measured as spectral power modifications (prevalence of electroencefalographic frequencies) between T0 and T1 and T1 and T2 | 1 to 2 years (2nd year)
  Significant outcome will be a shift of frequency band.
  A significant outcome will be a shift of frequency band.
Neuropsychological testing: improvement between T0 and T1 and T1 and T2. | 1 to 2 years (2nd year)
  Cut-off values cannot be defined a priori, and their range will be included into secondary endpoints.
Mean change in visual analogue scale (VAS) for pain | 1 to 2 years (2nd year)
  Changes in scores of VAS (pain perception) will be recorded
Mean change in Short Form (36) Health Survey for NP | 1 to 2 years (2nd year)
  Changes in scoresShort Form (36) Health Survey (perceived quality of life) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Del Felice, PhD, Principal Investigator — University of Padua, Italy
Locations (1):
- University Hospital, Padua, Italy

IPD SHARING:
Plan to Share IPD: Yes
Studdy protocol will be shared with any ORCID resgistered scientist at any time upon request
Supporting Information: Study Protocol
Access Criteria: ORCID Registered scientists at any time

REFERENCES:
- [Result] Del Felice A, Castiglia L, Formaggio E, Cattelan M, Scarpa B, Manganotti P, Tenconi E, Masiero S. Personalized transcranial alternating current stimulation (tACS) and physical therapy to treat motor and cognitive symptoms in Parkinson's disease: A randomized cross-over trial. Neuroimage Clin. 2019;22:101768. doi: 10.1016/j.nicl.2019.101768. Epub 2019 Mar 18. PMID 30921609